CLINICAL TRIAL: NCT06652568
Title: Determining the Validity of ThinkSono Guidance for Ultrasound Image Acquisition and Remote Detection
Acronym: DVT GUARD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ThinkSono, Ltd. (Industry)
Collaborators: NYU Langone Health (Other); Temple Health (Unknown); Allegheny Health Network (Other); University of Wisconsin, Madison (Other); South Texas Veterans Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 012023
Record Dates: First submitted 2024-10-12; First posted 2024-10-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Deep Vein Thrombosis; Deep Vein Thrombosis, Pulmonary Embolus
Keywords: Deep vein thrombosis; Artificial intelligence; Machine learning; Ultrasound
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Single arm comparison study between the ThinkSono device and standard of care venous duplex ultrasound.
Masking Description: Though not masked, the study is double blinded. Double blinding will be ensured by the ThinkSono software, as it will not be giving any indication of diagnosis or image quality to the operator. The comparison scan will be done by a qualified imaging specialist as per the standard of care at the local institution, but they will also not know the results of the ThinkSono scan. There will also be "remote qualified clinicians" reviewing the ThinkSono data (separately from local staff) who also will not know the results of the local imaging specialist. Only at the final data assessment upon study completion will outcome assessors be aware of ThinkSono device results and local site imaging results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Comparison Arm (Other): This arm of patients will undergo an ultrasound scan using the ThinkSono system and a comparison standard of care duplex ultrasound scan.
  Interventions: Device: ThinkSono System

INTERVENTIONS:
Device: ThinkSono System — The ThinkSono Guidance System is a guidance software expected to help non-radiology specialist healthcare professionals produce compression ultrasound image data that meet or exceed the minimal image quality criteria for a remote diagnosis by an expert (e.g. radiologist).

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of the ThinkSono Guidance System, a software data collection and communication tool designed to collect ultrasound data to help detect blood clots in veins. The ThinkSono system is CE Mark approved in the European Union and in clinical use in Europe. Usually, when an ultrasound is conducted to diagnose blood clots in veins, a sonographer (trained technologist who conducts ultrasounds) and/or radiologist will conduct the procedure, including a compression ultrasound exam, and the scan may require a bulky cart and ultrasound equipment. The ThinkSono Guidance System is a mobile software application that enables other healthcare professionals such as nurses, non-radiologist physicians including general practitioners, and other allied healthcare professionals to perform the ultrasound at the point of care using guidance from the software app. This is a multi-site non-randomized, double-blinded, prospective cohort pivotal study.

DETAILED DESCRIPTION:
Deep vein thrombosis (DVT) is well recognized to cause significant morbidity and mortality both at the time of diagnosis and post-diagnosis. With an estimated incidence of 1- 2 per 1,000 people, over to 300,000 people in the US will be diagnosed with venous thromboembolism (VTE) per annum and two-thirds of these will be DVT. However, positive cases only represent 12-25% of the total number of patients who present with suspected DVT. In other words, between 75-88% of suspected DVT cases, when fully investigated, are negative. Estimates have placed the yearly cost of VTE to the US healthcare system at up to $10 billion.

It is notoriously difficult to diagnose a DVT by clinical acumen alone. The standard approach to making a diagnosis of proximal DVT currently involves an algorithm combining pre-test probability assessment through the Well's score, and compression ultrasonography. Handheld ultrasound probes have recently become available. These probes have enabled 'app-based' compression ultrasonography to be performed without the need for bulky cart or laptop-based ultrasound machines. These new machines have a small form factor, meaning only the ultrasound probe is required for diagnostic purposes in conjunction with a smartphone or tablet.

At present, although the new handheld probes are smaller and are better suited for point of care diagnosis, they still require an experienced radiologist or sonographer to perform the compression exam. This means that these devices can only be used wherever sonographers/radiologists are based most often i.e. hospital radiology departments. However, due to recent advances in "machine learning", software is now being developed for these 'app-based' probes that can assist non-radiology specialist healthcare professionals (e.g. nurses, non-radiologist physicians, general practitioners and other allied healthcare professionals) to carry out the compression ultrasound exam with minimal training.

The ThinkSono Guidance System is a guidance software expected to help non-radiology specialist healthcare professionals produce compression ultrasound image data that meet or exceed the minimal image quality criteria for a remote diagnosis by an expert (e.g. radiologist). The ThinkSono system is CE Mark approved in the European Union and in clinical use in Europe.

This study is a multi-site non-randomized, double-blinded, prospective cohort pivotal study. The purpose of this study is to confirm the safety and efficacy of the ThinkSono Guidance System as per the intended use defined as:

ThinkSono Guidance System is a guidance, data acquisition and communication tool that guides non-ultrasound-trained healthcare staff to collect point of care compression ultrasound data in the proximal deep venous system of the lower extremity for interpretation by qualified clinicians.

ELIGIBILITY:
Inclusion Criteria:

* The participant is willing to provide written informed consent to participate in this research.
* The participant is over the age of 18
* The participant has symptoms suggestive of a deep venous thrombosis (DVT)
* The diagnostic DVT algorithm indicates that an ultrasound is needed

Exclusion Criteria:

* Patient consent not given or retracted during the study.
* Local imaging specialists fail to scan the patient or fail to produce a conclusive imaging diagnosis.
* Incomplete ThinkSono Guidance scan due to logistical or other issues such as pain, lack of patient cooperation, barriers such as a cast or other physical limitations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Image quality adequacy | Through study completion, an average of 8 months.
  At least 75% of the data collected by non-specialist operators of the study team via the ThinkSono Guidance App is adequate for interpretation (i.e., with an American College of Emergency Physicians (ACEP) score equal to or greater than 3) as rated by a remote qualified clinician.

SECONDARY OUTCOMES:
ThinkSono system sensitivity | Through study completion, an average of 8 months.
  Measure the sensitivity of the compressibility assessment in the proximal venous system by the remote qualified clinicians using data from the ThinkSono Guidance Mobile App compared against the assessment of the local imaging technologists using standard of care ultrasound.
ThinkSono system specificity | Through study completion, an average of 8 months.
  Measure the specificity of the compressibility assessment in the proximal venous system by the remote qualified clinicians using data from the ThinkSono Guidance Mobile App compared against the assessment of the local imaging technologists using standard of care ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Jacobowitz, MD, Principal Investigator — Northwell Health
Locations (5):
- United States (5):
  - NYU Langone Health, New York, New York
  - Temple Health, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - South Texas Veterans Health System, San Antonio, Texas
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nothnagel K, Aslam MF. Evaluating the benefits of machine learning for diagnosing deep vein thrombosis compared with gold standard ultrasound: a feasibility study. BJGP Open. 2025 Jan 2;8(4):BJGPO.2024.0057. doi: 10.3399/BJGPO.2024.0057. Print 2024 Dec. PMID 38866404
- [Background] Poulikidis KP, Gasparis AP, Labropoulos N. Prospective analysis of incidence, extent and chronicity of lower extremity venous thrombosis. Phlebology. 2014 Feb;29(1):37-42. doi: 10.1258/phleb.2012.012086. Epub 2013 May 6. PMID 23131597
- [Background] Grosse SD, Nelson RE, Nyarko KA, Richardson LC, Raskob GE. The economic burden of incident venous thromboembolism in the United States: A review of estimated attributable healthcare costs. Thromb Res. 2016 Jan;137:3-10. doi: 10.1016/j.thromres.2015.11.033. Epub 2015 Nov 24. PMID 26654719
- [Background] Prandoni P, Kahn SR. Post-thrombotic syndrome: prevalence, prognostication and need for progress. Br J Haematol. 2009 May;145(3):286-95. doi: 10.1111/j.1365-2141.2009.07601.x. Epub 2009 Feb 13. PMID 19222476
- [Background] Roberts LN, Patel RK, Donaldson N, Bonner L, Arya R. Post-thrombotic syndrome is an independent determinant of health-related quality of life following both first proximal and distal deep vein thrombosis. Haematologica. 2014 Mar;99(3):e41-3. doi: 10.3324/haematol.2013.089870. Epub 2014 Jan 17. No abstract available. PMID 24441147
- [Background] Kearon C, Julian JA, Newman TE, Ginsberg JS. Noninvasive diagnosis of deep venous thrombosis. McMaster Diagnostic Imaging Practice Guidelines Initiative. Ann Intern Med. 1998 Apr 15;128(8):663-77. doi: 10.7326/0003-4819-128-8-199804150-00011. PMID 9537941
- [Background] Kainz B, Heinrich MP, Makropoulos A, Oppenheimer J, Mandegaran R, Sankar S, Deane C, Mischkewitz S, Al-Noor F, Rawdin AC, Ruttloff A, Stevenson MD, Klein-Weigel P, Curry N. Non-invasive diagnosis of deep vein thrombosis from ultrasound imaging with machine learning. NPJ Digit Med. 2021 Sep 15;4(1):137. doi: 10.1038/s41746-021-00503-7. PMID 34526639
- [Background] Oppenheimer J, Mandegaran R, Staabs F, Adler A, Singohl S, Kainz B, Heinrich M, Geroulakos G, Spiliopoulos S, Avgerinos E. Remote Expert DVT Triaging of Novice-User Compression Sonography with AI-Guidance. Ann Vasc Surg. 2024 Feb;99:272-279. doi: 10.1016/j.avsg.2023.08.022. Epub 2023 Oct 10. PMID 37820986
- See also: Study sponsor website — http://thinksono.com